CLINICAL TRIAL: NCT04358172
Title: The Use of Mobile Application as a Tool for Patient Education
Brief Title: The Effectiveness of a Mobile Application in Educating Partial Denture Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Ho Ting Khee, Lecturer and Prosthodontist, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JEP-2018-583
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Mobile Applications
Keywords: Progressive web application, Denture care, Oral Hygiene

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated into the intervention group (educated using mobile application) and control group (educated using verbal instructions accompanied by demonstrations on dental models)
Who Masked: Outcomes Assessor
Masking Description: The clinician who check the oral index is masked with the group of subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app (Experimental): Participants in this group is educated using the mobile application
  Interventions: Other: 'Oral and Denture Guide' mobile application
- Control (No Intervention): Participants in this group is educated using the conventional method practised in the Faculty of Dentistry, National University of Malaysia (verbal instructions accompanied by demonstrations on dental models)

INTERVENTIONS:
Other: 'Oral and Denture Guide' mobile application — 'Oral and Denture Guide' mobile application provides evidence-based information about cleaning aids and material for dentures, denture care and oral hygiene instructions.
  Arms: Mobile app

SUMMARY:
A randomised control trial to evaluate the effect of a mobile application on partial denture wearers's dental knowledge, oral hygiene and denture hygiene. The null hypothesis of the study states that there will be no difference in dental knowledge, oral and denture hygiene among patients educated using the mobile application compared to those educated using the conventional method of verbal instructions accompanied by demonstrations on dental models.

DETAILED DESCRIPTION:
Partial denture wearers are at higher risk of developing caries and periodontal disease. Thus, providing oral and denture hygiene care instructions after denture delivery is crucial for prevention of oral diseases. A mobile application was developed using the progressive web application technology for chairside education and to serve as a reference material. The effect of the mobile application on patient's dental knowledge compared to the conventional method was evaluated using a knowledge questionnaire administered before and after education. The knowledge scores obtained were analysed using the Two-way mixed ANOVA test. Patients' oral hygiene was assessed by comparing the Silness and Loe Plaque Index and Gingival Index scores before and after education. Denture hygiene was evaluated by comparing the denture plaque score before and after education. Statistical analysis of the Plaque Index, Gingival Index and denture plaque score was done using Mann-Whitney U Test and Friedman Test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients wearing cobalt-chromium removable partial denture made in the dental laboratory in UKM and delivered by undergraduate students from June 2017 to June 2019 in the Faculty of Dentistry, National University of Malaysia.
2. Patients who own a smart phone with internet access and have been using it within the last six months.
3. Patients aged 25-75 years old.
4. Patients that are literate in English or Malay language.

Exclusion Criteria:

1. Patients who do not wear their removable partial dentures or only wear them occasionally.
2. Patients with a history of denture repair or reline, and those using denture adhesive.
3. Patients with physical or mental disabilities that will impede their ability to perform oral hygiene activities.
4. Patients involved in other oral-health education or oral hygiene maintenance program.
5. Patients who are active smokers.
6. Patients with medical conditions that may affect the gingival health, such as drug-induced gingival hypertrophy or Sjögren syndrome.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score | Change from baseline knowledge score at 3 months after education
  Participants' knowledge of oral and denture hygiene care. Minimum value:0, Maximum value:20. Higher score better

SECONDARY OUTCOMES:
Change in Plaque Index score | Change from baseline Plaque Index score at 1 month and 3 months after education
  Participants' oral hygiene
Change in Gingival Index score | Change form baseline Gingival Index score at 1 month and 3 months after education
  Participants' oral hygiene
Change in Denture plaque score | Change from baseline denture plaque score at 1 month and 3 months after education
  Participants' denture hygiene. Minimum value:0, Maximum value:4. Lower score better

CONTACTS AND LOCATIONS:
Overall Officials: Ting Khee Ho, MSc, Principal Investigator — National University of Malaysia
Locations (1):
- Faculty of Dentistry, National University of Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majchrzak, T. A., Biørn-Hansen, A. & Grønli, T.-M. 2018. Progressive Web Apps: the definite approach to cross-platform development? Proceedings of the 51st Hawaii International Conference on System Sciences, pp. 5735-5744.
- [Background] Zaror C, Espinoza-Espinoza G, Atala-Acevedo C, Munoz-Millan P, Li Y, Clarke K, Onetto J, Diaz J, Hallet K, Manton D, Marino R. Validation and usability of a mobile phone application for epidemiological surveillance of traumatic dental injuries. Dent Traumatol. 2019 Feb;35(1):33-40. doi: 10.1111/edt.12444. Epub 2018 Oct 25. PMID 30248238
- [Background] Nielsen, J. 1994. Heuristic evaluation. In Nielsen, J. & Mack (ed.). Usabiility Inspection Methods., pp. 25-62. New York: John Wiley and Sons.
- [Background] Sauro, J. & Lewis, J. R. 2016. Standardized usability questionnaires. Quantifying the User Experience, pp. 185-248. Elsevier Inc.
- [Background] Brooke, J. 1996. SUS-A quick and dirty usability scale. In Jordan, Patrick W.,Thomas, B. & Weerdmeester (ed.). Usability Evaluation in Industry, pp. 189-194. London: Taylor & Francis.
- [Background] Mohamad Marzuki MF, Yaacob NA, Yaacob NM. Translation, Cross-Cultural Adaptation, and Validation of the Malay Version of the System Usability Scale Questionnaire for the Assessment of Mobile Apps. JMIR Hum Factors. 2018 May 14;5(2):e10308. doi: 10.2196/10308. PMID 29759955
- [Background] Bujang, M. A. & Baharum, N. 2017. A simplified guide to determination of sample size requirements for estimating the value of intraclass correlation coefficient: A review. Archives of Orofacial Sciences The Journal of the School of Dental Sciences 12(1): 1-11.
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Augsburger RH, Elahi JM. Evaluation of seven proprietary denture cleansers. J Prosthet Dent. 1982 Apr;47(4):356-9. doi: 10.1016/s0022-3913(82)80079-6. No abstract available. PMID 6951034
- See also: Guide on how to built progressive web application — https://www.goodbarber.com/blog/progressive-web-apps-everything-you-need-to-know-a895/